CLINICAL TRIAL: NCT07362082
Title: A Randomized Clinical Trial of Telehealth Treatment for Opioid Use Disorders
Brief Title: A Clinical Trial of Telehealth Treatment for Opioid Use Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000041129; 4R33DA057675-02 (NIH); 1R61DA057675-01 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RecoveryPad platform (Experimental): Participants randomized to RecoveryPad platform
  Interventions: Device: RecoveryPad platform
- Treatment as usual (No Intervention): Treatment as usual: referrals to harm reduction and other community resources that are already being given to individuals in the various community and healthcare settings from which these participants are being recruited.

INTERVENTIONS:
Device: RecoveryPad platform — Telehealth platform to enhance motivation and engagement in treatment for OUD
  Arms: RecoveryPad platform

SUMMARY:
This trial will assess effects of enrollment in a comprehensive telehealth platform, RecoveryPad (RP), in adults with moderate or severe opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Can speak, read and write in English
* Provision of signed and dated informed consent form
* Screened positive for OUD, moderate or severe, based on the Diagnostic and Statistical Manual-5th Edition
* Have a working cell phone number and working device that can access a web browser and receive texts (i.e., smartphone, tablet or computer)
* Can provide a working email address OR be willing to create one

Exclusion Criteria:

* Current use of buprenorphine, methadone, or naltrexone for a substance use disorder
* Pregnancy or lactation
* Known current suicide risk based on participant self-report
* On parole or incarcerated at time of enrollment based on participant self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Mean time to first buprenorphine prescription | 30 days post enrollment
  Mean time to first buprenorphine prescription within 30 days of engagement with RP.

SECONDARY OUTCOMES:
Number of participants with current MOUD prescription | 90 days post enrollment
  Number of participants with a current prescription of MOUD at 90 days
Mean number overdose events | 30 and 90 days post enrollment
  Mean number of overdose events at 30 and 90 days
Number of participants with methadone referral and induction | 90 days post enrollment
  Number of participants with methadone referral and induction

CONTACTS AND LOCATIONS:
Overall Officials: Rebekah Heckmann, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes